CLINICAL TRIAL: NCT04617899
Title: The Study to Evaluate the Performance and Safety of the Novasight Hybrid System Using Objective Performance Criteria
Acronym: SUPERIOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CardioNavi MedTech (Wuhan) Co., Ltd. (Industry)
Collaborators: Beijing Jingruitianhe Medical Science and Technology Development Co,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CardioNavi
Record Dates: First submitted 2020-10-21; First posted 2020-11-05 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease
Keywords: Intravascular imaging; Intravascular ultrasound; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Novasight IVUS/OCT (Experimental): A coronary segment with stent will be imaged by the Novasight IVUS/OCT catheter
  Interventions: Diagnostic Test: Intravascular imaging

INTERVENTIONS:
Diagnostic Test: Intravascular imaging — Use of imaging catheter

SUMMARY:
This prospective, multicenter, single-arm study aims to evaluate the safety, operability and practicability of the novel hybrid intravascular imaging system/catheter during the percutaneous transluminal coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age and less than 85 years of age.
2. Subject must be informed and sign a written consent
3. Subject must have evidence of myocardial ischemia, unstable angina or acute myocardial infarction suitable for PCI.

Exclusion Criteria:

1. Women who are pregnant or cannot eliminate the possibility to be pregnant.
2. Estimated creatinine clearance <30 ml/min/1.73 m2 using Cockcroft equation.
3. LVEF(Left ventricular ejection fraction) < 35% by the most recent imaging test within 7 days prior to procedure.
4. Unstable ventricular arrhythmias.
5. High bleeding risk, active peptic ulcers or cerebrovascular accident or transient ischemic attack within the past 6 months.
6. Known contraindication to anticoagulants and antiplatelets therapy.
7. Known hypersensitivity to aspirin, clopidogrel, heparin, iodinated contrast, ticagrelor, bivalirudin, metal materials in stent.
8. Any intervention for not target vessel within 48 hours after the study procedure.
9. Any conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation.

Angiographic exclusion criteria:

1. The reference diameter of target vessel is less than 2.5 mm.
2. The target lesion involves myocardial bridge.
3. The target lesion is in the left main coronary artery or the damage is observed in the ostium.
4. Severe calcification in the target vessel.
5. Severe tortuosity in the target vessel.
6. Multiple contiguous stent implantation in the target vessel.
7. Subject has coronary artery spasm.
8. In-stent restenosis.
9. Any study lesion characteristic that, in the investigator's opinion, is not available for intravascular imaging.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clear image length measured by Core lab | During the procedure
  The clear image length is transformed from the clear image frame, and the ratio of the clear image can be calculated by Clear image length / Full image length * 100%

SECONDARY OUTCOMES:
Catheter-related major adverse events | Periprocedure
  Cardiac death, myocardial infarction, blood-limited dissection
Clear stent length measured by Core lab | During the procedure
  Clear stent length is defined as the total stent length visualized within the clear image length.
Device Success | During the procedure
  Successfully deliver the catheter to the target lesion and withdrawal without fracture
Technical Success | During the procedure
  Successfully imaging
Image quality evaluated by operator | During the procedure
  Objective and subjective assessment of image quality.
System reliability evaluated by operator | During the procedure
  Objective and subjective assessment of system reliability.
Catheter operability evaluated by operator | During the procedure
  Objective and subjective assessment of catheter operability.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Chaoyang District
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Fengtai District
  - Chinese PLA General Hospital, Beijing, Haidian District
  - Peking University Third Hospital, Beijing, Haidian District

IPD SHARING:
Plan to Share IPD: No
According to the policy of the Human Genetic Resource Administration of China, the data is limited and it could not be shared currently.

REFERENCES:
- [Derived] Jin Q, Fu Z, Wang Y, Zeng Y, Zhang X, Ye Y, Tang Y, Xu X, Chen Y. A Multicenter Feasibility and Safety Study of a Novel Hybrid IVUS-OCT Imaging System. JACC Asia. 2025 Mar;5(3 Pt 1):396-400. doi: 10.1016/j.jacasi.2025.01.009. PMID 40049934